CLINICAL TRIAL: NCT07212933
Title: The Safety and Clinical Efficacy of RAK Cell Therapy in Late-stage Gastric Cancer: A Randomized Controlled Trial
Acronym: RAK in GC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Lin Chen, Prof., Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S2025-443-02
Record Dates: First submitted 2025-10-02; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Gastric (Stomach) Cancer; Biological Therapy; Immunotherapy
Keywords: Gastric cancer; late-stage; progression-free survival; chemotherapy; T cell biological therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — trifluridine tipiracil drug combination; Trifluridine; tipiracil

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: A "double-dummy" method will be used. Based on the randomization results, the investigational drug (RAK cell suspension), TAS-102 (oral drug), and the infusion simulator (normal saline + small amount of fat emulsion) will have their outer packaging marked as either Group A or Group B drugs, making it indistinguishable which is the experimental or control group drug. However, different dosage forms within a group can be distinguished. Medical personnel unaware of the patient's drug group assignment will administer the Group A or Group B drugs to patients according to the corresponding sequence in the randomization table. Unblinding will occur at the end of the study follow-up or when necessary during the treatment process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAS-102+RAK cell (Experimental): Combined therapy of RAK cells and TAS-102
  Interventions: Biological: RetroNectin active Killer cells; Drug: TAS-102 (trifluridine and tipiracil, Lonsurf®)
- TAS-102 (Active Comparator): sole use of TAS-102
  Interventions: Drug: TAS-102 (trifluridine and tipiracil, Lonsurf®)

INTERVENTIONS:
Biological: RetroNectin active Killer cells — RetroNectin-Activated Killer (RAK) cells, derived from autologous peripheral blood mononuclear cells (PBMCs), are induced in vitro by RetroNectin along with anti-CD3 monoclonal antibody and Interleukin-2 (IL-2). These cells consist of various cytotoxic effectors, primarily CD8+ T (cytotoxic T, Tc) cells and natural killer T cells, which exhibit minimal cytotoxicity to normal cells but substantial specificity to tumor cells, thereby demonstrating both safety and potent anti-tumor activity.
  Arms: TAS-102+RAK cell
Drug: TAS-102 (trifluridine and tipiracil, Lonsurf®) — Based on the results of the RECOURSE [16] and TERRA [17] studies, TAS-102 (Trifluridine/Tipiracil Hydrochloride) will be administered orally at a dose of 35mg/m², twice daily, Days 1-5, with each cycle lasting 3 weeks.

SUMMARY:
This project employs a prospective, double-blind, randomized controlled trial methodology to comparatively analyze the safety and survival outcomes of human umbilical cord blood RAK cells applied in advanced gastric cancer. Firstly, the maximum tolerated dose (MTD) of RAK cell therapy for patients with advanced gastric cancer will be determined through a dose-escalation trial. Subsequently, the overall survival (OS), progression-free survival (PFS), and incidence of adverse events will be compared between the RAK treatment group and the control group. This aims to explore the efficacy and safety of biotherapy for recurrent or metastatic gastric cancer where frontline therapy has failed, thereby laying the foundation and providing evidence for large-scale, multi-center clinical studies.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects voluntarily join this study and sign the informed consent form. 2. Age ≥18 years and ≤70 years. 3. Confirmed by gastroscopic pathology or imaging (enhanced CT/PET-CT) as Stage IV gastric cancer or gastroesophageal junction adenocarcinoma (cTanyNanyM1). Metastatic sites include but are not limited to: liver, peritoneum, lungs, pancreas, greater omentum, retroperitoneal lymph nodes, etc.

  4. Failure or disease progression after prior frontline anti-tumor therapy (including ineffective first- and second-line chemotherapy, targeted therapy, and immunotherapy for advanced gastric cancer).

  5. Have measurable solid tumors (efficacy evaluation standard: RECIST 1.1); tumor assessment via CT scan or MRI must be performed within 28 days before treatment.

  6. Physical performance status ECOG 0-3. 7. Expected lifespan ≥1 month. 8. Participants must be able to understand the study procedures and agree to participate in the study by providing written informed consent.

Exclusion Criteria:

* 1. Concurrent other types of malignancy. 2. Severe cardiac, pulmonary, or cerebral system diseases. 3. Expected survival <1 month. 4. Laboratory investigations indicating unsuitability for receiving anti-tumor biotherapy:

  1. Moderate to severe bone marrow suppression: (HGB <80 g/L; WBC <2.0×10⁹/L; ANC <1.0×10⁹/L; PLT <50×10⁹/L).
  2. Significantly decreased liver function (Child-Pugh Grade C).
  3. Severe renal insufficiency (CKD Stage III and above).
  4. Severe coagulation dysfunction (INR ≥1.5 or APTT >1.5 × ULN).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | one-year
  Progression-Free Survival (PFS) is the length of time during and after treatment that a patient's cancer does not get worse. It measures how long the disease remains stable or in remission.

SECONDARY OUTCOMES:
Overall Survival | one-year
  from a defined randomization until death from any cause.
Objective Response Rate (ORR) | one-year
  the proportion of patients in a clinical trial whose cancer shrinks (responds) by a predefined amount for a minimum period of time. It is a direct measure of a drug's anti-tumor activity.
Time to Progression (TTP) | one-year
  the length of time from the start of treatment (or randomization in a trial) until the patient's cancer is objectively documented to have worsened.

OTHER OUTCOMES:
Biotherapy-related adverse reactions | one-year
  side effects caused by a class of cancer treatments known as Biological Therapies: Dermatitis: Skin rash and itching.
  Hepatitis: Inflammation of the liver, detected by elevated liver enzymes in blood tests.
  Pneumonitis: Inflammation of the lungs, causing cough, shortness of breath, and chest pain. This can be life-threatening.
  Endocrinopathies: Inflammation of hormone glands, leading to conditions like:
  Thyroiditis (underactive or overactive thyroid).
  Hypophysitis (inflammation of the pituitary gland).
  Adrenal Insufficiency (where the body can't manage stress).
  Less Common but Serious: Can affect almost any organ, including the heart (myocarditis), muscles (myositis), kidneys (nephritis), and nervous system (neuropathy).
Blood immunology indicators | one-year
  T-cell count, IL-2/IL-6/IL-11, TGF-β,

CONTACTS AND LOCATIONS:
Locations (1):
- The First＆Fifth Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The ethics committee which approved this study required the individual participante should be anoymization.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-30): https://cdn.clinicaltrials.gov/large-docs/33/NCT07212933/Prot_SAP_000.pdf